CLINICAL TRIAL: NCT03132324
Title: A Phase 1 Open-Label, Dose-Escalation Study to Evaluate Safety, Pharmacokinetic, and Biological Activity of INCB059872 in Subjects With Sickle Cell Disease
Brief Title: A Study to Evaluate Safety, Pharmacokinetic, and Biological Activity of INCB059872 in Subjects With Sickle Cell Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study is terminated due to a business decision not to pursue INCB059782 in Sickle Cell Disease indication.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 59872-102
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease (SCD); sickle cell SS; lysine demethylase 1 (LSD1) inhibition
MeSH Terms: conditions — Anemia, Sickle Cell; Inhibition, Psychological | interventions — INCB059872

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- INCB059872 0.5 mg (Experimental): INCB059872 0.5 mg tablet administered orally every other day (QOD) for 28 days on an empty stomach. If dose was well tolerated, once daily (QD) administration was evaluated independently and in parallel with QOD administration.
  Interventions: Drug: INCB059872
- INCB059872 1 mg (Experimental): INCB059872 1 mg tablet administered orally QOD for 28 days on an empty stomach. If dose was well tolerated, QD administration was evaluated independently and in parallel with QOD administration.
  Interventions: Drug: INCB059872
- INCB059872 2 mg (Experimental): INCB059872 2 mg tablet administered orally QOD for 28 days on an empty stomach. If dose was well tolerated, QD administration was evaluated independently and in parallel with QOD administration.
  Interventions: Drug: INCB059872

INTERVENTIONS:
Drug: INCB059872 — INCB059872 tablets

SUMMARY:
The purpose of this study was to evaluate the safety and tolerability, and the pharmacokinetic and biologic activity of INCB059872 in participants with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCD (sickle cell SS) confirmed through hemoglobin electrophoresis.
* Must be red blood cell (RBC) transfusion-independent (not currently on regularly scheduled transfusions) for ≥ 3 months from the time of first dose of study drug.
* No RBC transfusion within 30 days of first dose of study drug.
* Hydroxyurea (HU) refractory

  -Must not have received HU therapy during the 3 months before receiving study drug.
* Creatinine clearance ≥ 60 mL/min based on the institutional formula.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Any unresolved toxicity ≥ Grade 2 from previous therapy except for stable chronic toxicities not expected to resolve.
* Pregnant or nursing women or participants expecting to conceive or father children within the projected duration of the study, starting with screening visit through completion of safety follow-up.
* Received an investigational study drug within 28 days or 5 half-lives (whichever is longer) before receiving the first dose of study drug (requirement may be waived with medical monitor approval).
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment.
* Prior receipt of LSD1 inhibitor therapy for any indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of INCB059872 assessed by monitoring frequency, duration, and severity of adverse events | Screening through 35 days after end of treatment, up to approximately 3 months per participant.
  An adverse event is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent.
Change in fetal hemoglobin (HbF) from baseline | Baseline through 2 weeks after end of treatment, up to approximately 2.5 months per participant.
  Pharmacodynamic activity assessed by measuring changes of HbF from baseline and their correlation to INCB059872 treatment. The HbF (F cells) in human whole blood will be characterized using flow cytometry.

SECONDARY OUTCOMES:
Cmax of INCB059872 | Baseline to Day 28.
  Defined as maximum observed plasma concentration.
AUC0-t of INCB059872 | Baseline to Day 28.
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Fitzroy Dawkins, MD, Study Director — Incyte Corporation
Locations (7):
- United States (7):
  - Acevedo Clinical Research Associates, Miami, Florida
  - Advanced Pharma, Miami, Florida
  - Vita Health and Medical Center, Tamarac, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Boston University, Boston, Massachusetts
  - Virginia Commonwealth University, Richmond, Virginia
  - Blood Centers of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No